CLINICAL TRIAL: NCT04074902
Title: Role of Chest Sonography in Evaluation of Successful Pleurodesis in Patients With Malignant Pleural Effusion
Brief Title: Role of Chest Sonography in Evaluation of Pleurodesis in Patients With Malignant Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Ahmed EL-Sagheir Adam, Principal investigator, Assiut University
Other Study IDs: Ultrasaund after pleurodesis
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Pleurodesis
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonography — Mindray dp1100 plus.

SUMMARY:
Thoracic ultrasonography easily detects the movement of the visceral pleura on the parietal pleura This sign is absent when pleurodesis is successful.

DETAILED DESCRIPTION:
Malignant pleural effusion (MPE) imposes a significant burden on patients and health-care providers. Most of the malignant pleural effusions are the result of metastases to the pleura from other sites. The primary tumors were, in the decreasing order of frequency: lung (37%), breast (17%), unknown site (10%), lymphoma (9%), gastrointestinal (8%), ovary (7%) and mesothelioma (3%) .

Management of malignant effusions depends on palliation of dyspnea and prevention of the re accumulation of pleural fluid to provide the highest possible quality of life, regardless of the need for other treatment modalities. Most patients require definitive treatment, usually drainage and chemical pleurodesis to relieve symptoms and prevent fluid recurrence. Pleurodesis is defined as the symphysis between the visceral and parietal pleural surfaces; its function is to prevent accumulation of either air or fluid into the pleural space. Effusions of malignant origin are the most common indication for pleurodesis Thoracic ultrasound (TUS) can easily visualize pleural effusions and help in identifying malignant effusion and the presence of pleural adhesions or thick pleural peel and could therefore have a role in predicting long-term pleurodesis success or failure in MPE.

One of the easiest sign to identify during chest sonography is the movement of the visceral pleura compared to immobility of the parietal pleura. This sign of 'pleural sliding', firstly described in veterinary medicine and was used to exclude the presence of pneumothorax when present and to suspect atelectasis, fibrosis or pleural adhesions (pleurodesis) when absent. Thoracic ultrasonography easily detects the sign of 'pleural sliding', due to the movement of the visceral pleura on the parietal pleura This sign is absent when pleurodesis is successful. Contrast-enhanced chest CT has become the imaging modality of choice to detect pleural effusions and assist the differentiation between benign andmalignant effusions detected bystandard radiographs. Chest CT findings characteristic of malignant pleural disease include (i) circumferential pleural thickening, (ii) nodular pleural thickening, (iii) parietal pleural thickening greater than 1 cm, and (iv) mediastinal pleural involvement or evidence of a primary tumour.(9'10) The reported specificities of each of these individual findings range from 22% to 56% and sensitivities range from 88% to 100%.(9;11) Histological confirmation of the diagnosis, however, remains necessary. Chest CT should be performed before large-volume thoracocentesis to allow visualization of both the visceral and parietal pleurae, which may identify a pleural mass and appropriate site for needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with malignant pleural effusion who will undergo palliative treatment with insertion of intercostal tube.

Exclusion Criteria:

1. Patients <18 years old, unable to provide informed consent.
2. Had an allergy or other contraindication to intrapleural pleurodesis.
3. Had evidence of unexpandable lung believed by the responsible clinician to represent insufficient.
4. pleural apposition that would preclude pleurodesis, and/or had an expected survival of<1 month.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients will be chosen at random for one year from the start of the study and will be recruited from chest out patient clinc and department Assiut University hospital which are eligible for this study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate and compare the outcome of pleurodisis by different modalities. | baseline
  To compare chest sonographic findings versus Multislice CT findings in detecting endobronchial obstruction in patients with malignant pleural effusion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corcoran JP, Hallifax RJ, Mercer RM, Yousuf A, Asciak R, Hassan M, Piotrowska HE, Psallidas I, Rahman NM. Thoracic Ultrasound as an Early Predictor of Pleurodesis Success in Malignant Pleural Effusion. Chest. 2018 Nov;154(5):1115-1120. doi: 10.1016/j.chest.2018.08.1031. Epub 2018 Sep 20. PMID 30243566